CLINICAL TRIAL: NCT04190797
Title: Photobiomodulation on Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Marcia Uchoa Rezende, Full Professor in Orthopedics and Traumatology, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23338619.4.0000.0068
Record Dates: First submitted 2019-12-03; First posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Knee Osteoarthritis; Metabolic Disease
Keywords: Laser Therapy; Osteoarthritis; Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Metabolic Diseases; Osteoarthritis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Photobiomodulation + patiente controled anaethesia (PCA) group (G1): patients in the immediate postoperateve of knee arthroplasty surgery treated with the Photobiomodulation device connected, 24h and 48h after the peripheral nerve block (femoral nerve and obturator nerve). With conventional analgesia and with the device of PCA.
  Interventions: Device: Photobiomodulation + patiente controled anaethesia (PCA)
- Control (Active Comparator): Placebo + PCA group (G2): patients undergoing knee arthroplasty surgery treated with the Photobiomodulation device switched off, in 24h and 48h after peripheral nerve blockade (femoral nerve and obturator nerve). With conventional analgesia and with the PCA apparatus.
  Interventions: Device: Placebo + patiente controled anaethesia (PCA)

INTERVENTIONS:
Device: Photobiomodulation + patiente controled anaethesia (PCA) — Patients in the immediate postoperateve of knee arthroplasty surgery treated with the Photobiomodulation device connected, 24h and 48h after the peripheral nerve block (femoral nerve and obturator nerve). With conventional analgesia and with the device of PCA.
  Arms: Experimental
Device: Placebo + patiente controled anaethesia (PCA) — Patients in the immediate postoperateve of knee arthroplasty surgery treated with the Photobiomodulation device switched off, in 24h and 48h after peripheral nerve bloc (femoral nerve and obturator nerve). With conventional analgesia and with the device of PCA.
  Arms: Control

SUMMARY:
Objective: This study is designed to evaluate the short-term efficacy of photobiomodulation for improving pain and function in patients that will undergo total knee replacement and decrease in morphine consumption and adverse effects of opioids. Methods: thirty four patients of both genders that will undergo total knee replacement will participate in this randomized controlled double-blind clinical trial. They will be randomly allocated into two groups: Photobiomodulation group 1 with 18 patients and placebo group with 18 patients and group 3 control without device . Photobiomodulation will be performed twice during 48h, using adivice Light-Aid da BrightPhotomedicine- Brasil, com LED de Arsenieto, Gálio and Alumínio (AsGaAl) of 850 nm device 3B class, measured and calibrated previously .Five points were irradiated on the knee. The placebo group will be treated with the same laser device, but will not be turned on. All patients will receive treatment sessions of photobiomodulation after 24h and 48 h after peripheral nerve blockade (femoral nerve block and nerve supply), applied in 5 points for 5 minutes (300 seconds) close to the incision (that will be protected by transparent film) and repeated every 24h after totaling 2 applications. Patients will be assessed for duration of surgery and anesthesia, assessment of the pain, time to first rescue analgesia request, physical examination, dosimetry of photobiomodulation and amount of morphine consumption using PCA 24h and 48 hours after nerve blockade after surgery. In addition, adverse effects , sedation, paresthesias, motor blockade, nausea and vomiting will be assessed ever 6h during 48h.

DETAILED DESCRIPTION:
thirty-four patients treated at the Institute of Orthopedics and Traumatology, University of São Paulo School of Medicine Hospital das Clínicas (IOT-HC-FMUSP), already identified with knee OA awaiting TKA; the thirty-four selected patients will be divided into two groups with 17 patients in each group:

* Photobiomodulation + PCA Group (G1): patients in the PO of knee arthroplasty surgery treated with the photobiomodulation device turned on, 24h and 48h after peripheral nerve block (femoral nerve and obturator nerve) .With conventional analgesia and with the device of PCA.
* Placebo + PCA group (G2): patients in the postoperative period of knee arthroplasty surgery treated with the photobiomodulation device switched off at 24h and 48h after peripheral nerve block (femoral nerve and obturator nerve). With conventional analgesia and with the PCA device.

All patients will undergo photobiomodulation treatment sessions after 24h and 48h of peripheral nerve block (femoral and adductor nerve block), applied in two regions: in the femoral nerve region for 4 minutes (240 seconds) and near the surgical incision (protected with clear film) for 2 minutes (120 seconds) and repeated every 24 hours after, totaling 2 applications in 2 regions (see table 1). Patients will be systematically evaluated with identification, duration of surgery and duration of anesthesia, pain assessment, time of first analgesic rescue request, physical examination, photobiomodulation dosimetry and amount of PCA bolus requested every 6h within within 48 hours after nerve block after knee arthroplasty surgery. In addition to assessing and quantifying adverse effects (motor block, sedation, nausea and vomiting). All pain assessments (VAS) and rescue number requests will be performed by "blinded examiners", ie professionals who will not be aware of the group to which the patient will belong.

ELIGIBILITY:
Inclusion Criteria:

* Men and women diagnosed with OAJ with comorbidities (metabolic syndrome, ie, OAJ + at least two overweight / central obesity, diabetes, dyslipidemia, high blood pressure)
* Age between 60 and 75 years awaiting primary TKA at IOT-HC-FMUSP
* Patients not submitted to previous lower limb arthroplasty.
* Patients not submitted to knee infiltration up to 6 months before study.
* Patients without personal history of cognitive, psychiatric and / or neurological disorders, whose symptoms presented at the moment of the evaluation are related or significantly interfere with the functions of attention, memory, logical reasoning, understanding, in order to impair the assimilation of the given guidelines.
* Patients with no personal history of inflammatory arthritis (rheumatoid arthritis, for example)

Exclusion Criteria:

* Contraindication for spinal anesthesia and / or peripheral nerve block
* Not having consent signed
* Prior use of strong opioids
* Unable to use PCA method
* Patients undergoing knee infiltration during the study.
* Patients diagnosed with chronic inflammatory arthritis (rheumatoid arthritis, for example) during the study.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate if photobiomodulation improves postoperative pain by VAS during hospital stay. | Day 2 after procedure
  Apply the VAS (Visual Analog Scale), range: 0 no pain - 100 worse pain

SECONDARY OUTCOMES:
Evaluate adverse events arising within 48 hours after surgery | Day 2 after procedure
  Will evaluate at 6:00 (immediate postoperative day) 6:00 , 12:00., 18:00 (1st postoperative day) and 6:00 and 12:00 (second postoperative day)
Evaluate morphine consumption in a patient-controlled analgesia device (PCA) from the immediate postoperative period up to 48h after the procedure | Day 2 after procedure
  Through the patient-controlled analgesia (PCA) method
Measure time to first request for analgesia rescue after peripheral nerve block | Day 2 after procedure
  Through the patient-controlled analgesia (PCA) method

CONTACTS AND LOCATIONS:
Overall Officials: George Freire, MD, Principal Investigator — University of São Paulo General Hospital

REFERENCES:
- [Background] Hawker GA, Badley EM, Borkhoff CM, Croxford R, Davis AM, Dunn S, Gignac MA, Jaglal SB, Kreder HJ, Sale JE. Which patients are most likely to benefit from total joint arthroplasty? Arthritis Rheum. 2013 May;65(5):1243-52. doi: 10.1002/art.37901. PMID 23459843
- [Background] Fedriani de Matos JJ, Atienza Carrasco FJ, Diaz Crespo J, Moreno Martin A, Tatsidis Tatsidis P, Torres Morera LM. Effectiveness and safety of continuous ultrasound-guided femoral nerve block versus epidural analgesia after total knee arthroplasty. Rev Esp Anestesiol Reanim. 2017 Feb;64(2):79-85. doi: 10.1016/j.redar.2016.05.008. Epub 2016 Jul 9. English, Spanish. PMID 27400891
- [Background] Gan TJ, Habib AS, Miller TE, White W, Apfelbaum JL. Incidence, patient satisfaction, and perceptions of post-surgical pain: results from a US national survey. Curr Med Res Opin. 2014 Jan;30(1):149-60. doi: 10.1185/03007995.2013.860019. Epub 2013 Nov 15. PMID 24237004
- [Background] Pogatzki-Zahn EM, Segelcke D, Schug SA. Postoperative pain-from mechanisms to treatment. Pain Rep. 2017 Mar 15;2(2):e588. doi: 10.1097/PR9.0000000000000588. eCollection 2017 Mar. PMID 29392204
- [Background] Shanthanna H, Huilgol M, Manivackam VK, Maniar A. Comparative study of ultrasound-guided continuous femoral nerve blockade with continuous epidural analgesia for pain relief following total knee replacement. Indian J Anaesth. 2012 May;56(3):270-5. doi: 10.4103/0019-5049.98776. PMID 22923827
- [Background] Al-Zahrani T, Doais KS, Aljassir F, Alshaygy I, Albishi W, Terkawi AS. Randomized clinical trial of continuous femoral nerve block combined with sciatic nerve block versus epidural analgesia for unilateral total knee arthroplasty. J Arthroplasty. 2015 Jan;30(1):149-54. doi: 10.1016/j.arth.2014.07.032. Epub 2014 Jul 31. PMID 25149364
- [Background] Karu T. Primary and secondary mechanisms of action of visible to near-IR radiation on cells. J Photochem Photobiol B. 1999 Mar;49(1):1-17. doi: 10.1016/S1011-1344(98)00219-X. PMID 10365442
- [Background] Pinto FC, Chavantes MC, Pinto NC, Alho EJ, Yoshimura EM, Matushita H, Krebs VL, Teixeira MJ. Novel treatment immediately after myelomeningocele repair applying low-level laser therapy in newborns: a pilot study. Pediatr Neurosurg. 2010;46(4):249-54. doi: 10.1159/000319363. Epub 2010 Dec 15. PMID 21160232
- [Background] Bjordal JM, Ljunggren AE, Klovning A, Slordal L. Non-steroidal anti-inflammatory drugs, including cyclo-oxygenase-2 inhibitors, in osteoarthritic knee pain: meta-analysis of randomised placebo controlled trials. BMJ. 2004 Dec 4;329(7478):1317. doi: 10.1136/bmj.38273.626655.63. Epub 2004 Nov 23. PMID 15561731
- [Background] Tam G. Low power laser therapy and analgesic action. J Clin Laser Med Surg. 1999 Feb;17(1):29-33. doi: 10.1089/clm.1999.17.29. PMID 10204446
- [Background] Masoumipoor M, Jameie SB, Janzadeh A, Nasirinezhad F, Soleimani M, Kerdary M. Effects of 660- and 980-nm low-level laser therapy on neuropathic pain relief following chronic constriction injury in rat sciatic nerve. Lasers Med Sci. 2014 Sep;29(5):1593-8. doi: 10.1007/s10103-014-1552-1. Epub 2014 Mar 16. PMID 24634001
- [Background] Medalha CC, Di Gangi GC, Barbosa CB, Fernandes M, Aguiar O, Faloppa F, Leite VM, Renno AC. Low-level laser therapy improves repair following complete resection of the sciatic nerve in rats. Lasers Med Sci. 2012 May;27(3):629-35. doi: 10.1007/s10103-011-1008-9. Epub 2011 Oct 19. PMID 22009383
- [Background] Fukuda VO, Fukuda TY, Guimaraes M, Shiwa S, de Lima Bdel C, Martins RA, Casarotto RA, Alfredo PP, Bjordal JM, Fucs PM. SHORT-TERM EFFICACY OF LOW-LEVEL LASER THERAPY IN PATIENTS WITH KNEE OSTEOARTHRITIS: A RANDOMIZED PLACEBO-CONTROLLED, DOUBLE-BLIND CLINICAL TRIAL. Rev Bras Ortop. 2015 Dec 6;46(5):526-33. doi: 10.1016/S2255-4971(15)30407-9. eCollection 2011 Sep-Oct. PMID 27027049
- [Derived] de Rezende MU, Varone BB, Martuscelli DF, Ocampos GP, Freire GMG, Pinto NC, de Sousa MVP. Pilot study of the effect of therapeutic photobiomodulation on postoperative pain in knee arthroplasty. Braz J Anesthesiol. 2022 Jan-Feb;72(1):159-161. doi: 10.1016/j.bjane.2021.07.040. Epub 2021 Nov 17. PMID 34800495